CLINICAL TRIAL: NCT05497297
Title: An Open-label, Single-dose Study to Assess the Pharmacokinetics of HSK7653 Tablets in Subjects With Varying Degrees of Renal Impairment Compared to the Control Subjects With Normal Renal Function
Brief Title: A Study to Evaluate the Pharmacokinetics of HSK7653 in Subjects With Renal Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Haisco Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSK7653-106
Record Dates: First submitted 2022-08-09; First posted 2022-08-11 (Actual); Last update posted 2023-01-03 (Actual); Status verified 2022-08

CONDITIONS: Renal Impairment
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Mild Renal Impairment (Experimental): A1 group subjects will receive a single dose of 10 mg HSK7653
  Interventions: Drug: HSK7653 tablets
- Moderate Renal Impairment (Experimental): B1 group subjects will receive a single dose of 10 mg HSK7653
  Interventions: Drug: HSK7653 tablets
- Severe Renal Impairment (Experimental): C1 group subjects will receive a single dose of 10 mg HSK7653
  Interventions: Drug: HSK7653 tablets
- Kidney failure (Experimental): D1 group subjects will receive a single dose of 10 mg HSK7653
  Interventions: Drug: HSK7653 tablets
- Normal Renal function (Experimental): A2, B2, C2 and D2 group subjects will receive a single dose of 10 mg HSK7653, If the age, sex and weight of the subjects in group A2 can be matched with the subjects in groups A1 and B1 at the same time, the subjects in group B2 will not be enrolled, and so on.
  Interventions: Drug: HSK7653 tablets

INTERVENTIONS:
Drug: HSK7653 tablets — HSK7653, tablet, oral
  Other Names: HSK7653

SUMMARY:
This is an open-label, single-dose study to evaluate the pharmacokinetics, pharmacodynamics and safety of HSK7653 in subjects with mild, moderate, severe renal impairment and subjects with kidney failure compared to the matched control subjects with normal renal function.

DETAILED DESCRIPTION:
This is an open-label, single-dose Phase I study that evaluate the pharmacokinetics, pharmacodynamics and safety of a single dose of HSK7653 10 mg in subjects with mild, moderate, and severe renal impairment , subjects with kidney failure and the control subjects with normal renal function. This study consists of a screening period (Day -14 to Day -1), a baseline period (Day -1), a treatment period (Day 1 to Day 29), and a follow-up call on Day 32.

Subjects will be enrolled in the following groups:

Glomerular filtration rate (GFR, unit mL/min/1.73m^2) will be calculated based on Modification of Diet in Renal Disease (MDRD) equation at screening, Multiply it by BSA, then divide by 1.73 to convert to absolute GFR (unit, mL/min) (group A1) mild renal impairment (60 ≤ GFR< 90 mL/min); (group B1) moderate renal impairment (30 ≤ GFR<60 mL/min); (group C1) severe renal impairment (15 ≤ GFR< 30 mL/min); (group D1) kidney failure (<15 mL/min, not on hemodialysis); (group A2,B2,C2,D2) control subjects with normal renal function will be matched with subjects with renal impairment by weight, age, and sex (GFR≥90 mL/min).If subjects in group A2 can be matched with the subjects in groups A1 and B1 at the same time, the subjects in group B2 will not be enrolled, and so on.

Approximately 64 subjects will be enrolled in total.

ELIGIBILITY:
Inclusion Criteria:

Subjects with renal impairment(RI):

1. Voluntarily sign the informed consent form, understand the trial procedures, and be willing to comply with all trial procedures and restrictions;
2. 18 years to 79 years (inclusive), male and female;
3. Male subjects weight ≥50 kg and female subjects weight ≥45 kg. Body mass index (BMI) : 18-30 kg/m2 (inclusive) (BMI= weight (kg)/height2 (m^2));
4. Subjects with medically stable RI until study completion corresponding to the Classifications of Renal Function based on GFR: mild RI: 60≤GFR<90 mL/min; moderate RI: 30≤GFR<60 mL/min, severe RI:15≤GFR<30 mL/min, kidney failure:GFR<15 mL/min (not on hemodialysis);
5. Physical examination, vital sign measurements, 12-lead electrocardiogram (ECG), and clinical laboratory tests (hematology, serum chemistry, coagulation and urinalysis test) results were deemed appropriate by the investigator;
6. Not in use of any drug within 2 weeks prior to screening, except for the medication necessary for RI/ other comorbidities (last more than four weeks in good compliance);
7. Subjects (including partners) are willing to voluntarily use effective contraceptives from screening to at least 6 months after the last dose administration;

Subjects with normal renal function :

1. Voluntarily sign the informed consent form, understand the trial procedures, and be willing to comply with all trial procedures and restrictions;
2. 18 years to 79 years (inclusive), male and female, age and sex must be matched with subjects with RI;
3. Male subjects weight ≥50 kg and female subjects weight ≥45 kg, weight must be matched with subjects with RI. Body mass index (BMI) : 18-30 kg/m^2 (inclusive) (BMI= weight (kg)/height2 (m^2));
4. 90≤GFR<130 mL/min;
5. Physical examination, vital sign measurements, 12-lead electrocardiogram (ECG), and clinical laboratory tests (hematology, serum chemistry, coagulation and urinalysis test) results were deemed appropriate by the investigator;
6. Not in use of any drug within 2 weeks prior to screening, except for the medication necessary for comorbidities (last more than four weeks in good compliance);
7. Subjects (including partners) are willing to voluntarily use effective contraceptives from screening to at least 6 months after the last dose administration；

Exclusion Criteria:

1. Subjects who have a allergic history of DPP4 inhibitors or have a history of allergy to the test drug and the related compounds;
2. Have a history of severe and uncontrolled diseases, such as cardiovascular, respiratory, liver, gastrointestinal, endocrine, hematologic, mental/nervous systems diseases within one year prior to screening；
3. History or clinical evidence of acute or chronic pancreatitis, or clinically significant abnormalities in blood lipase and/or blood amylase results at screening;
4. Have conditions that may affect drug absorption, distribution, metabolism, or excretion (e.g., disease, drugs or surgery);
5. Use of any DPP-IV enzyme inhibitor within 2 weeks prior to the screening;
6. Experienced severe hypoglycemia within 3 months before screening;
7. Acute renal failure;
8. Smoking more than 5 cigarettes per day within 3 months prior to screening or smoking during the study；
9. Average alcohol intake is more than 14 unit per week (1unit=17.7 mL alcohol , 1 unit=357mL 5% alcohol beer, or 43mL 40% alcohol spirit, or 147mL 12% alcohol wine) within the 3 months prior to screening, or taking any alcohol during study or a positive ethanol breath test at screening;
10. Drug abuse history within 5 years prior to screening, or positive urine drug screen at screening；
11. History of high consumption of grapefruit juice, methylxanthine-rich food or beverage (such as coffee, tea, cola, chocolate, energy drinks) , consumption of grapefruit juice, methylxanthine-rich food within 48 hours before the administration ；
12. Participation in another clinical trial within 3 months before screening；
13. Blood donation (or blood loss) ≥400 mL, or receiving blood products to improve anemia within 3 months prior to the screening；
14. Aspartate aminotransferase (AST), alanine aminotransferase (ALT) > 2 × upper limit of normal, or bilirubin > 1.5 × upper limit of normal；
15. Have a positive result for hepatitis B surface antigen, hepatitis C virus antibody, human immunodeficiency virus antibody, or anti-treponema pallidum specific antibody；
16. A pregnant/lactating woman, or has a positive pregnancy test at screening or during the trial；
17. Not suitable for this study as judged by the investigator.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2022-08-04 (Actual); Primary Completion 2022-10-23 (Actual); Study Completion 2022-10-26 (Actual)

PRIMARY OUTCOMES:
Cmax | Predose and 0.25, 0.5, 1, 2, 4, 8 , 12, 24, 72, 168, 336, 504, 672 hours after dosing
  The pharmacokinetic parameters of HSK7653 in plasma
AUC0-t | Predose and 0.25, 0.5, 1, 2, 4, 8 , 12, 24, 72, 168, 336, 504, 672 hours after dosing
  The pharmacokinetic parameters of HSK7653 in plasma
AUC0-inf | Predose and 0.25, 0.5, 1, 2, 4, 8 , 12, 24, 72, 168, 336, 504, 672 hours after dosing
  The pharmacokinetic parameters of HSK7653 in plasma

SECONDARY OUTCOMES:
Tmax | Predose and 0.25, 0.5, 1, 2, 4, 8 , 12, 24, 72, 168, 336, 504, 672 hours after dosing
  The pharmacokinetic parameters of HSK7653 in plasma
t1/2 | Predose and 0.25, 0.5, 1, 2, 4, 8 , 12, 24, 72, 168, 336, 504, 672 hours after dosing
  The pharmacokinetic parameters of HSK7653 in plasma
Vz/F | Predose and 0.25, 0.5, 1, 2, 4, 8 , 12, 24, 72, 168, 336, 504, 672 hours after dosing
  The pharmacokinetic parameters of HSK7653 in plasma
CL/F | Predose and 0.25, 0.5, 1, 2, 4, 8 , 12, 24, 72, 168, 336, 504, 672 hours after dosing
  The pharmacokinetic parameters of HSK7653 in plasma
Ae | Predose and 168 hours after dosing
  The pharmacokinetic parameters of HSK7653 in urine
Fe | Predose and 168 hours after dosing
  The pharmacokinetic parameters of HSK7653 in urine
CLr | Predose and 168 hours after dosing
  The pharmacokinetic parameters of HSK7653 in urine
DPP4 inhibition AUEC | Predose and 1, 24, 72, 168, 336 hours after dosing
  The pharmacodynamic parameters of HSK7653 in plasma
DPP4 inhibition Emax | Predose and 1, 24, 72, 168, 336 hours after dosing
  The pharmacodynamic parameters of HSK7653 in plasma
DPP4 inhibition E336h | Predose and 1, 24, 72, 168, 336 hours after dosing
  The pharmacodynamic parameters of HSK7653 in plasma
The number of volunteers with adverse events as a measure of safety | Day 1 to Day 32
  The number of volunteers with adverse events as a measure of safety

CONTACTS AND LOCATIONS:
Overall Officials: Wang Meixia, Principal Investigator — Beijing Jishuitan Hospital; Zhang dongliang, Principal Investigator — Beijing Jishuitan Hospital
Locations (1):
- Beijing Jishuitan Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shi D, Chen L, Li G, Wu N, Zhang F, Wang X, Mu N, Chen X, Yang X, Lu J, Lu Y, Wang M, Zhang D. Pharmacokinetics, Pharmacodynamics, and Safety of Single Dose HSK7653 Tablets in Chinese Subjects with Normal or Impaired Renal Function. Clin Pharmacokinet. 2024 Feb;63(2):227-239. doi: 10.1007/s40262-023-01333-4. Epub 2024 Jan 6. PMID 38184489